CLINICAL TRIAL: NCT05438160
Title: A Multi-center, Exploratory, Single-Arm, 7-week Study to Evaluate the Feasibility and Acceptability of the Medication Tracking and Educational Components of a Clinical Learning Version of CT-155 in People With Schizophrenia
Brief Title: Exploratory Study of a Digital Therapeutics in People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Click Therapeutics, Inc. (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CT-155-C-003
Record Dates: First submitted 2022-05-18; First posted 2022-06-29 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
Keywords: Prescription digital therapeutics; Smartphone app; Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Clinical Learning Study version of CT-155 (Other): Single arm acceptability and feasibility of medication tracking and educational components of a clinical learning study version of CT-155
  Interventions: Device: Clinical Learning Study smartphone app (i.e., the study app)

INTERVENTIONS:
Device: Clinical Learning Study smartphone app (i.e., the study app) — The study app is designed to provide 7-weeks of the medication tracking and educational components in a clinical learning study version of CT-155. This design allows inferences to be made about the usability and acceptability of these components of CT-155. Eligible participants will be enrolled during an in-person clinic visit on Day 1. Participants will then be directed to access the study app and perform tasks each day for the 49-day engagement period.

SUMMARY:
CT-155 is a novel prescription digital therapeutic (PDT) being developed by Click Therapeutics, Inc. (Click) and Boehringer Ingelheim (BI) using an interactive, software-based intervention to treat schizophrenia

DETAILED DESCRIPTION:
CT-155 is a novel prescription digital therapeutic (PDT) being developed by Click Therapeutics, Inc. (Click) and Boehringer Ingelheim (BI). CT-155 delivers an interactive, software-based intervention for schizophrenia.

This is a multi-center, exploratory, single-arm study to evaluate the feasibility and acceptability of medication tracking and educational component of a clinical learning study version of CT-155 in adults diagnosed with schizophrenia.

Eligible participants must have a diagnosis of schizophrenia per Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5).

Participants that meet eligibility criteria will be enrolled in the study on Day 1. The study consists of an up to 7-day screening period, a 49-day engagement period, and an up to 7-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* 1. Is willing and able to provide written informed consent to participate in the study, attend study visits, and comply with study-related requirements and assessments.
* 2. Between 18 and 64 years of age at time of informed consent.
* 3. Fluent in written and spoken English, confirmed by ability to read and understand the informed consent form.
* 4. Has a primary diagnosis of schizophrenia using the diagnostic criteria for schizophrenia as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5), for at least 1-year prior to screening.
* 5. Is in the stable phase of illness, as assessed by the investigator after review of medical records or documented discussion with the treating physician.
* 6. Has outpatient treatment status at the time of screening, with no inpatient treatment for schizophrenia within 12 weeks prior to screening.
* 7. Is on a stable dose of antipsychotic medication(s) for at least 12 weeks prior to enrollment (Day 1) as determined by the investigator.
* 8. Has obtained a score of 30 or less on the MAP-SR as assessed at the screening visit.
* 9. Is the sole user, per participant self-report, of an iPhone with an iPhone operating system (iOS) 13 or greater or a smartphone with an Android operating system 9 or greater and is willing to download and use the Study App as required per the protocol.
* 10. Is the owner of, and has regular access to, an email address.
* 11. Has regular access to the internet via cellular data plan and/or wifi.
* 12. Has stable housing and has remained at the same residence for at least 12 weeks prior to screening, with no anticipated housing changes during the duration of the study.
* 13. Understands how to use the Study App during the screening visit as assessed by the investigator during in-clinic Study App installation and activation activities.

Exclusion Criteria:

* 1. Is currently treated with more than two antipsychotic medications (including more than two dosage forms).
* 2. Is currently treated with clozapine or haloperidol.
* 3. Has active prominent positive symptoms in the opinion of the investigator that would preclude effective engagement in treatment for negative symptoms.
* 4. Is currently receiving or has received psychotherapy within 12 weeks prior to screening.
* 5. Meets either the International Classification of Diseases, Tenth Revision (ICD-10) or DSM-5 criteria for diagnoses not under investigation, including schizophreniform, schizoaffective, or psychosis non-specific disorders.
* 6. Has post-traumatic stress disorder (PTSD), bipolar disorder, major depressive disorder, developmental disorders, or any prominent disorder that would interfere with compliance to the protocol, per investigator judgment.
* 7. Has substance or alcohol use disorder (excluding caffeine and nicotine), that would interfere with compliance to the protocol, per investigator judgment.
* 8. Currently needs or will likely require prohibited concomitant medications and/or therapy during the study, as determined by the investigator.
* 9. Is currently participating in another clinical study (interventional or observational) involving investigational drugs or devices.
* 10. Prior participation in the CT-155-C-001 clinical study.
* 11. Has suicidal ideation or behavior, as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS):

  1. Participants with a "yes" response to either Items 4 or 5 on the C-SSRS Suicidal Ideation Item within the last 12 weeks prior to screening or at baseline visit.
  2. Participants with a "yes" response on the C-SSRS Suicidal Behavior Items within the last 26 weeks prior to screening or at baseline visit.
  3. Participants who, in the opinion of the investigator, present a serious risk of suicide.
* 12. In the judgment of the investigator, any evidence of a clinically significant concomitant disease or any other clinical condition that would jeopardize the participant's safety while participating in the clinical study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
To explore feasibility and acceptability of the medication tracking and educational components of a clinical learning study version of the CT-155 app | Day 49 at the end of treatment period
  Degree of participant engagement with the study app as measured by participant app use data captured in-app

SECONDARY OUTCOMES:
Change from Week 3 of the Mobile Agnew Relationships Measure | Change from Week 3 to Week 7 of the Mobile Agnew Relationships Measure
  To explore the establishment of a digital working alliance over the course of the Study as assessed by the change from Week 3 to Week 7 of the Mobile Agnew Relationships Measure.
  The Mobile Agnew Relationships Measures is on a 7-item scale that ranges from "Strongly Disagree" as scale 1 to "Strongly Agree" as scale 7.

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Lakhan, MDPhD, FAAN, Study Chair — Click Therapeutics
Locations (7):
- United States (7):
  - CT-155 Center, Anaheim, California
  - CT-155 Center, Torrance, California
  - CT-155 Center, Hialeah, Florida
  - CT-155 Center, Lake Mary, Florida
  - CT-155 Center, Miami, Florida
  - CT-155 Center, Irving, Texas
  - CT-155 Center, Richmond, Texas

IPD SHARING:
Plan to Share IPD: No